CLINICAL TRIAL: NCT07134114
Title: Comparative Evaluation of Occlusal Changes Following Hall Technique Crowns in Different Primary Molar Groups: A Randomized Controlled Clinical Trial
Brief Title: Occlusal Impact of Hall Crowns in Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, AYŞE IŞIL CİHAN, Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-25-11969
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Dental Occlusion; Pediatric Dentistry
Keywords: Hall technique; Occlusal adjustment; Intraoral scanning
MeSH Terms: conditions — Dental Caries; Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The biostatistician performing the data analysis will be blinded to group allocation. The clinician performing treatment and model analysis will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maxillary First Primary Molar (Experimental): A preformed metal crown will be placed and cemented on the carious maxillary first primary molar using the Hall Technique, without any tooth preparation or administration of local anesthesia.
  Interventions: Procedure: Hall Technique
- Maxillary Second Primary Molar (Active Comparator): A preformed metal crown will be placed and cemented on the carious maxillary second primary molar using the Hall Technique, without any tooth preparation or administration of local anesthesia.
  Interventions: Procedure: Hall Technique
- Mandibular First Primary Molar (Active Comparator): A preformed metal crown will be placed and cemented on the carious mandibular first primary molar using the Hall Technique, without any tooth preparation or administration of local anesthesia.
  Interventions: Procedure: Hall Technique
- Mandibular Second Primary Molar (Active Comparator): A preformed metal crown will be placed and cemented on the carious mandibular second primary molar using the Hall Technique, without any tooth preparation or administration of local anesthesia.
  Interventions: Procedure: Hall Technique

INTERVENTIONS:
Procedure: Hall Technique — Procedure: Hall Technique A preformed stainless-steel crown will be placed on a primary molar using the Hall Technique. This approach does not require local anesthesia, caries removal, or tooth preparation.
  Digital Scan and Bite Registration Schedule:
  * T0 (Baseline): Immediately before crown placement
  * T1 (Immediate): Immediately after crown placement
  * T2 (Two Weeks): Two weeks after crown placement
  * T3 (One Month): One month after crown placement At each time point (T0-T3), digital scans of both the upper and lower arches will be obtained, and a bite registration will be recorded. These records will be used to generate three-dimensional digital models, which will be analyzed to assess occlusal relationships and monitor changes over time.

SUMMARY:
Hall Technique is a non-invasive restorative approach for managing carious primary molars, increasingly used in pediatric dentistry due to its simplicity and patient tolerance. This study aims to evaluate and compare the occlusal changes that occur following Hall crown placement on different primary molar groups (maxillary first molar, maxillary second molar, mandibular first molar, mandibular second molar) using digital model analysis.

DETAILED DESCRIPTION:
The aim of this clinical study is:

* to evaluate the occlusal changes that occur following the Hall Technique in different primary molar groups.
* to investigate whether the molar group (first vs. second) and jaw location (maxilla vs. mandible) influence the degree or pattern of occlusal adaptation.

A total of 60 healthy children aged between 7 and 10 years will be recruited from the Pediatric Dentistry Clinic at Ankara Yıldırım Beyazıt University, Faculty of Dentistry. Patients must have at least two primary molars requiring restorative treatment and meet all inclusion criteria.

After obtaining informed consent from parents and assent from the child, one eligible primary molar per participant will be randomly selected for Hall crown placement using a computer-generated allocation system. Based on the selected tooth, participants will be stratified into four groups: Group 1 (Maxillary first primary molar), Group 2 (Maxillary second primary molar), Group 3 (Mandibular first primary molar), and Group 4 (Mandibular second primary molar). Following group allocation, all other necessary dental treatments-including conventional restorations, endodontic procedures, and preventive interventions-will be completed to eliminate potential occlusal interferences.

One week after the completion of all dental treatments other than the Hall Technique, a baseline digital intraoral scan will be obtained using the Trios 3 scanner (3Shape, Copenhagen, Denmark), prior to crown placement on the designated primary molar. The Hall Technique will then be applied without local anesthesia or any caries removal. Debris will be gently cleared from the cavity, and airway protection will be ensured using gauze or elastoplast fixation. An appropriately sized preformed stainless-steel crown will be filled with glass ionomer cement (3M Ketac Cem) and seated on the tooth. The child will be instructed to bite firmly to ensure crown placement, or finger pressure will be used if necessary. Excess cement will be removed and interproximal contacts will be cleaned with dental floss. Digital intraoral scans will be repeated at three additional time points: immediately after crown placement (T1), at two weeks (T2), and at one month (T3) post-treatment. Superimposition and occlusal analysis will be conducted using Trios CAD (Computer-Aided Design) software to evaluate changes in occlusal parameters over time.

Following parameters will be quantitatively assessed:

* Positional change (in mm) between the mesiobuccal, distobuccal, mesiolingual/palatal, and distolingual/palatal cusp tips of the Hall-treated tooth, as well as the cusp tips of the opposing teeth in maximum intercuspation with this tooth.
* Positional change (in mm) of the cusp tip of the maxillary primary canine on the same side as the treated tooth
* Positional change (in mm) between the mesiobuccal cusp tips of all permanent first molars,
* Change in anterior occluso-vertical dimension (in mm)
* Change in posterior occluso-vertical dimension (in mm)
* Change (in mm²) in the surface area of maximum occlusal contact regions, based on digital bite registration records.

Statistical analysis will involve comparing changes in linear (mm) and surface area (mm²) measurements across the four study groups at multiple time intervals (T0-T1, T0-T2, T0-T3, T1-T2, T1-T3, and T2-T3). Data distribution will be assessed using the Shapiro-Wilk test. Group comparisons will be performed using ANOVA, Kruskal-Wallis, chi-square, and two-way mixed ANOVA or F1-LD-F1 design, as appropriate. Bonferroni correction will be applied for post hoc tests, and p ≤ 0.05 will be considered statistically significant. Analyses will be conducted using SPSS v.23 and R software.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Participants

* No skeletal or dental anomalies,
* ASA (American Society of Anesthesiologists) physical status classification of I or II ,
* Frankl Behavior Rating Scale score of 3 or 4,
* In the mixed dentition stage,
* Fully erupted permanent first molars in occlusal contact at maximum intercuspation
* No acute dental pain or need for emergency treatment,
* Presence of at least two primary molars with carious lesions scored as 3, 4, or 5 according to the ICDAS (International Caries Detection and Assessment System),
* Presence of an antagonist tooth for the molar planned to receive Hall Technique,
* Provision of verbal and written informed consent by the participant and legal guardian after reading or listening to the consent form and fully understanding its content.

Inclusion Criteria for Tooth

Based on Clinical Examination:

* No history of prolonged pain in response to thermal or chemical stimuli, or spontaneous pain suggestive of irreversible pulpitis,
* No sensitivity to percussion or palpation,
* Absence of both pathological and physiological mobility,
* No signs of swelling, fistula, or discoloration,
* Sufficient remaining tooth structure to retain a preformed stainless steel crown.

Based on Radiographic Examination:

* Radiolucent lesion associated with dental caries located within the outer one-third to two-thirds of the dentin, with a visible band of normal dentin between the lesion and the pulp,
* At least two-thirds of root length present,
* No signs of internal or external pathological or physiological root resorption,
* Intact lamina dura and normal periodontal ligament space,
* No periradicular bone loss surrounding the roots,
* No calcified masses in the pulp chamber.

Exclusion Criteria:

* Individuals with serious systemic or psychological conditions
* Participants who fail to attend follow-up appointments
* Those who exhibit excessive fear or anxiety reactions and are unable to cooperate during treatment

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Cusp Tip Displacement (Linear Measurement in mm): | From Hall crown placement to 1 month after treatment completion
  The positional changes of the mesiobuccal, distobuccal, mesiolingual/palatal, and distolingual/palatal cusp tips of the crowned primary molar, as well as the cusp tips of the opposing teeth in maximum intercuspation with this tooth, will be measured by comparing the distances between each cusp tip across time points: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement).
Vertical Positional Change of the Maxillary Primary Canine Cusp Tip (Linear Measurement in mm) | From Hall crown placement to 1 month after treatment completion
  The vertical distance of the cusp tip of the maxillary primary canine located on the same side as the treated tooth will be measured at each time point: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement). The measurements will be compared within the same tooth across time points to assess any vertical displacement over time.
Vertical Positional Change of the Mesiobuccal Cusp Tips of All Permanent First Molars (Linear Measurement in mm) | From Hall crown placement to 1 month after treatment completion
  The vertical positions of the mesiobuccal cusp tips of all permanent first molars will be measured at each time point: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement). Intra-tooth comparisons will be performed to evaluate any vertical changes over time.
Anterior Occlusal Vertical Dimension (Linear Measurement in mm) | From Hall crown placement to 1 month after treatment completion
  The anterior occlusal vertical dimension will be assessed by measuring the vertical distance between the cusp tip of the maxillary primary canine and the cusp tip of the mandibular primary or permanent canine on the same side as the treated tooth. This measurement will be performed in maximum intercuspation at all time points: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement). If the mandibular primary or permanent canine on the same side is not present or cannot be measured, the corresponding canine on the contralateral side will be used.
Posterior Occlusal Vertical Dimension (Linear Measurement in mm) | From Hall crown placement to 1 month after treatment completion
  The posterior occlusal vertical dimension will be evaluated by measuring the vertical distance between the mesiobuccal cusp tips of the opposing maxillary and mandibular permanent first molars on the same side as the treated tooth. This measurement will be taken in maximum intercuspation at all time points: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement).
Change in Maximum Occlusal Contact Area (mm²) | From Hall crown placement to 1 month after treatment completion
  The change in maximum occlusal contact areas (in mm²) will be analyzed based on bite registration records. Since the Trios 3 software does not allow direct quantitative measurement of occlusal contact areas, the analysis will be performed using the color-coded occlusal contact maps generated by the software. Specifically, the red zones representing the areas of maximum contact will be identified from the screenshots, and their surface areas will be measured using the ImageJ software. This analysis will be two-dimensional, based on calibrated screenshots, and will provide a comparative assessment of occlusal contact area changes across different time points: T0 (immediately before crown placement), T1 (immediately after crown placement), T2 (two weeks after crown placement), and T3 (one month after crown placement).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe I. Cihan, Professor, Study Chair — Ankara Yıldırım Beyazit University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Dentistry, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akyildiz BM, Al-Yaseen W, Innes N, Zhurov A, Tas A, Sonmez I. Longitudinal observational digital analysis of occlusion in Hall Technique. J Dent. 2025 Feb;153:105547. doi: 10.1016/j.jdent.2024.105547. Epub 2024 Dec 30. PMID 39743130
- [Background] Joseph RM, Rao AP, Srikant N, Karuna YM, Nayak AP. Evaluation of Changes in the Occlusion and Occlusal Vertical Dimension in Children Following the Placement of Preformed Metal Crowns Using the Hall Technique. J Clin Pediatr Dent. 2020;44(2):130-134. doi: 10.17796/1053-4625-44.2.12. PMID 32271658
- [Background] Kaya MS, Kinay Taran P, Bakkal M. Temporomandibular dysfunction assessment in children treated with the Hall Technique: A pilot study. Int J Paediatr Dent. 2020 Jul;30(4):429-435. doi: 10.1111/ipd.12620. Epub 2020 Feb 12. PMID 31991506
- [Background] Gallagher S, O'Connell BC, O'Connell AC. Assessment of occlusion after placement of stainless steel crowns in children - a pilot study. J Oral Rehabil. 2014 Oct;41(10):730-6. doi: 10.1111/joor.12196. Epub 2014 Jun 10. PMID 24913609
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395